CLINICAL TRIAL: NCT03620357
Title: Continuous Glucose Monitoring & Management In Type 2 Diabetes
Brief Title: Continuous Glucose Monitoring & Management In Type 2 Diabetes (T2D)
Acronym: COMMITED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTL903076
Record Dates: First submitted 2018-07-31; First posted 2018-08-08 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, multicenter, two-arm pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Continuous Glucose Monitor (CGM) Group (Experimental)
  Interventions: Device: CGM
- SMBG Group (Active Comparator)
  Interventions: Device: SMBG

INTERVENTIONS:
Device: CGM — CGM Group: Dexcom G6 CGM
  Arms: Continuous Glucose Monitor (CGM) Group
Device: SMBG — SMBG Group: Blood Glucose Meter
  Arms: SMBG Group

SUMMARY:
A Study to assess if patients with Type 2 diabetes (T2D) who have suboptimal glycemic control using multiple oral agents are able to make lifestyle changes resulting in improved glycemic control by use of real-time continuous glucose monitoring (RT-CGM) and targeted learning modules versus self monitored blood glucose (SMBG) testing.

DETAILED DESCRIPTION:
The study is referred to as "Continuous Glucose Monitoring and Management in Type 2 Diabetes" also known as The COMMITED Study" and will assess if patients with Type 2 diabetes (T2D) who have suboptimal glycemic control using 2 or more multiple oral agents are able to make lifestyle changes resulting in improved glycemic control by use of real-time continuous glucose monitoring and targeted learning modules.

At time of enrollment, participants will undergo a run-in period of blinded CGM for a duration of 10 days to collect baseline data. Baseline Patient Report Outcome (PRO) surveys will be administered at the start of run-in.

The study design includes a run-in phase, a study phase and a follow up visit. During the study phase, participants will be randomized into two groups - CGM Group or SMBG Group. For the RT-CGM Group, the study comprises of 4 scheduled clinic visits at baseline (after Run-In), week 4, week 8, and week 12 to collect data on episodic RT-CGM use. During these visits, RT-CGM insertions will take place at baseline, week 4 and week 8 clinic visits, with each wear period lasting a duration of 10 days. For the SMBG Group, the study comprises of 3 scheduled clinic visits at baseline (after Run-In), week 8 (to collect data on episodic blinded CGM use) and week 12. CGM insertions will take place at week 8 with a wear period of 10 days. Both groups will have HbA1c collected at week 0 and week 12. The same PRO surveys administered at start of run-in will be administered again at week 12. There will not be therapeutic changes during the study phase unless needed for safety.

There will be phone/remote visits by a study site clinician at weeks 2, 6 and 10 in both groups to review the SMBG or CGM data. During these remote visits, there will be discussions about what the subjects have learned from their glucose monitoring and what the study clinician has observed.

All subjects will be scheduled for a follow up visit at Month 9 to obtain local lab or POC HbA1c. Diabetes medications (classifications only) will also be collected.

ELIGIBILITY:
Major Inclusion Criteria:

* Age at least 30 years
* Diagnosis of T2D treated with 2 or more oral anti-diabetic medications
* HbA1c ≥ 7.8 and ≤10.5% by local lab or POC

Major Exclusion Criteria:

* Using insulin
* Pregnancy
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
HbA1c | From baseline to Month 3 (Week 12)
  The primary endpoint is defined as change in HbA1c (determined by local lab or POC results).

CONTACTS AND LOCATIONS:
Overall Officials: David Price, MD, Study Director — DexCom, Inc.
Locations (10):
- United States (9):
  - Diabetes/Lipid Management and Research Center, Huntington Beach, California
  - Temecula Valley Endocrinology, Temecula, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - MODEL Clinical Research (Towson), Baltimore, Maryland
  - Diabetes & Endocrine Associates, PC, Omaha, Nebraska
  - Las Vegas Endocrinology, Henderson, Nevada
  - The Docs, Las Vegas, Nevada
  - Palm Research Center, Las Vegas, Nevada
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas
- LMC Manna Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No